CLINICAL TRIAL: NCT04292197
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled, Single/Multiple Day Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of 18- Methoxycoronaridine (18-MC HCl) Administered Orally to Normal Healthy Volunteers
Brief Title: A Study to Assess 18-Methoxycoronaridine (18-MC HCl) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Definium Therapeutics US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: MMED003
Record Dates: First submitted 2020-02-18; First posted 2020-03-03 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Addiction
Keywords: opioid use disorder (OUD)
MeSH Terms: conditions — Behavior, Addictive; Opioid-Related Disorders | interventions — 18-methoxycoronaridine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 18-MC SAD Study (Experimental): In Part 1, healthy participants will be randomized into cohorts to receive 18-MC HCl or placebo twice in 1 day.
  Interventions: Drug: 18-MC Compound
- 18-MC MAD Study (Experimental): In Part 2, healthy participants will be randomized into cohorts to receive 18-MC HCl or placebo twice a day for 7 consecutive days.
  Interventions: Drug: 18-MC Compound

INTERVENTIONS:
Drug: 18-MC Compound — 18-MC

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of a single day dosing and a separate multiple day dosing of 18-MC HCl administered orally, each part of the study having a different set of healthy male and female volunteers.

DETAILED DESCRIPTION:
This is a Phase 1, double-blind, randomized, placebo-controlled, single day and multiple day dosing, in healthy, non-smoking, male and female volunteers.

Part 1: Single Ascending Dose (SAD)

Seven (7) healthy male and female volunteers will be randomly assigned to receive either 18-MC HCl (n=5) or placebo (n=2) in each cohort. These volunteers will receive 18-MC HCl twice in 1 day (bid).

There are 3 phases: Screening, Enrollment and Follow-Up. All participants will be assessed for safety and tolerability for 28 days. Screening begins when a participant reports to the clinical unit (CU) for a screening visit to undergo safety and compliance assessments on this day. Participants that meet all eligibility criteria will be admitted to the CU on the day prior to receiving study drug. Enrollment begins on Day 1 where participants will receive two doses of study drug for 1 day, will be assessed for 18-MC PK up to 48 hours, and will remain admitted at the CU until Day 3, at which time they will be discharged. For follow-up the participants will return for safety and tolerability assessments at Days 7, 14, 21 and Day 28.

Part 2: Multiple Day Ascending Dose (MAD)

Seven (7) healthy male and female volunteers will be randomly assigned to receive either 18-MC HCl (n=5) or placebo (n=2) in each cohort. These volunteers will receive 18-MC HCl twice over 7 days (bid).

There are 3 phases: Screening, Enrollment and Follow-Up. All participants will be assessed for 42 days. Screening begins when a participant reports to the clinical unit (CU) for a screening visit to undergo safety and compliance assessments on this day. Participants that meet all eligibility criteria will be admitted to the CU on the day prior to receiving study drug. Enrollment begins on Day 1 where participants will receive two doses of study drug every day for 7 days, will be assessed for 18-MC PK up to 48 hours on Day 1 and Day 7, and will remain admitted at the CU until Day 9, at which time they will be discharged. For follow-up the participants will return for safety and tolerability assessments at Days 14, 21, 28, 35 and Day 42.

ELIGIBILITY:
Key Inclusion Criteria:

1. Written informed consent before any study-specific procedures.
2. Healthy male and female volunteers aged 18 to 55 years (inclusive) with suitable veins for cannulation and repeated venipuncture.
3. Female subjects of both childbearing and nonchildbearing potential will be considered, with certain conditions met
4. Female subjects must agree not to breastfeed starting at screening and throughout the study period.
5. Male participants must agree to practice abstinence; be surgically sterilized; or agree to use of a condom, plus effective contraception.
6. Have not smoked or used any tobacco or nicotine-containing products in the 3 months before screening and agree not to smoke during the entire study.

Key Exclusion Criteria:

1. History of any clinically important disease or disorder that, in the opinion of the investigator, would affect the ability of the participant to participate in the study
2. History or presence of gastrointestinal, hepatic, cardiac, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of study drug.
3. History of gastrointestinal ulcer disease, inflammatory bowel disease, or frequent indigestion symptoms
4. Adequate organ function
5. History of seizures or epilepsy.
6. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV).
7. Any clinically significant cardiovascular abnormalities
8. Known or suspected history of substance abuse disorder
9. History of alcohol abuse or excessive intake of alcohol
10. Positive screen for drugs of abuse, cotinine (nicotine) or alcohol
11. Has received another new chemical entity (defined as a compound, which has not been approved for marketing) or has participated in any other clinical study that included drug treatment within 30 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
To assess the safety, using incidence and severity of adverse events, of a single and multiple-day dosing of 18-MC administered orally. | Up to 28 days (SAD) and 42 days (MAD)
  Safety and tolerability will be assessed by the incidence and severity of adverse events (AEs). An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-SAEs.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 48 post dose - Day 1 and Day 7
  Blood samples for determination of study drug (18-MC) concentration parameters at various timepoints
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 48 hours post dose - Day 1 and Day 7
  Blood samples for determination of study drug (18-MC) parameters at various timepoints
Area Under the Curve from Time Zero to Last Quantifiable Concentration (AUClast) | AUC(t0-48hr) pg*hr/mL
  Blood samples for determination of study drug (18-MC) parameters at various timepoints
Terminal Elimination Half-Life (t1/2) | 48 hours post dose - Day 1 and Day 7
  Blood samples for determination of study drug (18-MC) concentration parameters at various timepoints
As an exploratory objective, the concentration of metabolites in plasma and urine may be determined | Up to 28 days (SAD) and 42 days (MAD)
  Plasma and urine samples for determination of study drug concentrations at various timepoints

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Sam Salman, Perth, Australia